Status: Effective 



Title

# Clinical Evaluation of a Silicone Hydrogel Daily Wear Monthly Replacement Contact Lens

Protocol Number: CLY935-C012 / NCT04422990

Development Stage of

Sponsor Name and

Project:

Development

Alcon Research, LLC and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Test Product: LID018869

Property of Alcon
Confidential
May not be used, divulged, published, or otherwise disclosed without the consent of
Alcon

Status: Effective 

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, all applicable regulatory authority regulations, and conditions of approval imposed by the reviewing IRB or regulatory authority.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's Brochure, product information, or other sources provided by the Sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements of the Sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you | ever been disqualified as an Investigator by any Regu | latory Authority? |
|---|---|---|---|
| | □ No | □Yes | |
| | Have you | ever been involved in a study or other research that w | as terminated? |
| | □ No | □Yes | |
| | If yes, ple | ase explain here: | |
| Pri | incipal Inve | estigator: | |
| | | Signature | Date |
| | ime and pro<br>sition: | ofessional | |
| Αċ | ldress: | | |

**Document:** TDOC-0057524 **Status:** Effective

Version: 1.0; CURRENT; Most-Recent; Effective


| | | <b>Table of Contents</b> | |
|----|-------------|------------------------------|----|
| Ta | ble of Co | ontents | 3 |
| Li | st of Table | es | 5 |
| Li | st of Figu | ires | 6 |
| 1 | GLOSS | ARY OF TERMS | |
| 2 | LIST O | F ACRONYMS AND ABBREVIATIONS | 11 |
| 3 | PROTO | OCOL SUMMARY | 13 |
| 5 | INTRO | DUCTION | 23 |
| | 5.1 | Rationale and Background | 23 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 25 |
| | 6.1 | Primary Objective(s) | 25 |
| | 6.2 | Secondary Objective(s) | 25 |
| | 6.4 | Safety Objective(s) | 26 |
| 7 | INVEST | TIGATIONAL PLAN | 26 |
| | 7.1 | Study Design | 26 |
| 0 | | | |
| 8 | | POPULATION | |
| | 8.1 | Inclusion Criteria | |
| | 8.2 | Exclusion Criteria | |
| Λ | 8.3 | Rescreening of Subjects | |
| 9 | | MENTS ADMINISTERED | |
| | 9.1 | Investigational Product(s) | 31 |

| Do | cument: TD | OC-0057524 Version: 1.0; CURRENT; Most-Recent; Effect | |
|---|---|---|---|
| Sta | tus: Effect | | Page <b>4</b> of <b>62</b> |
| | 9.3 | Treatment Assignment/Randomization | 36 |
| | 9.4 | Treatment masking | |
| | 9.5 | Accountability Procedures | 39 |
| | 9.6 | Changes to concomitant medications, treatments/ procedure | s39 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | 40 |
| | 10.1 | Informed Consent and Screening | 41 |
| | 10.2 | Description of Study Procedures and Assessments | 41 |
| | | 10.2.1 Demographics | 41 |
| | | 10.2.2 Medical History and Concomitant Medications | 41 |
| | | 10.2.3 Investigational Product compliance | 41 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 42 |
| | | 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment | |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 42 |
| | | 10.2.7 Visual Acuity: Effectiveness Assessment | 42 |
| | 10.5 | Discontinued Subjects | 43 |
| | | 10.5.1 Screen Failures | |
| | | 10.5.2 Discontinuations | |
| | | 10.5.3 Schedule of Procedures and Assessments for Subj<br>from Investigational Product | |
| | 10.6 | Clinical Study Termination | 44 |
| | | 10.6.1 Follow-up of subjects after study participation has | s ended45 |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 45 |
| | 11.1 | General Information | 45 |
| | 11.2 | Monitoring for AEs | 48 |
| | 11.3 | Procedures for Recording and Reporting | 48 |
| | 11.5 | Unmasking of the Study Treatment | 51 |
| | 11.6 | Follow-Up of Subjects with AEs | 51 |
| | 11.7 | Pregnancy in the Clinical Study | 51 |
| 12 | ANALY | SIS PLAN | |
| | 12.1 | Subject Evaluability | |
| | | Analysis Sets | |

| Alcon - Bus<br>Document: TD | | • | Version: 1.0; CURRENT; | Most-Recent; | | ite: 20-May-2020 |
|---|---|---|---|---|---|---|
| Status: Effect | | | v ersion. | | | Page <b>5</b> of <b>62</b> |
| | 12.2.1 | Safety A | nalysis Set | | | 52 |
| | 12.2.2 | Full Ana | lysis Set | | | 52 |
| | 12.2.3 | Per Prote | ocol Analysis Set | | | 53 |
| 12.3 | Demogra | aphic and | Baseline Characteristic | es | | 53 |
| 12.4 | Effective | eness Anal | lyses | | | 53 |
| | 12.4.1 | Analysis | of Primary Effectiven | ess Endpoint | (s) | 53 |
| | | 12.4.1.1 | Statistical Hypotheses | S | | 53 |
| | | 12.4.1.2 | Analysis Methods | | | 54 |
| | 12.4.2 | Analysis | of Secondary Effectiv | eness Endpo | ints | 54 |
| | | 12.4.2.1 | Statistical Hypotheses | S | | 54 |
| | | 12.4.2.2 | Analysis Methods | | | 54 |
| 12.6 | Safety A | nalyses | | | | 56 |
| 13 DATA H | ANDLING | G AND A | DMINISTRATIVE RE | QUIREMEN | TS | 57 |
| 13.1 | | | iality | | | |
| 13.2 | | | arce Documents and Ca | | | |
| 13.3 | | | Clarifications | | | |
| | | | toring Responsibilities | | | |
| 13.5 | | | nentation and Records | | | |
| 13.6 | | | and Quality Control | | | |
| | = | | und Quanty Control | | | |
| 14 ETHICS | | | | | ••••• | 00 |
| | | | List of Tables | 1 | | |

| | ness ese only | List of Figures List of Figures Current; Most-Recent; Effective Date: 26-May-2020 Additional content of the second of the sec |
|---|---|---|
| Document: TDC Status: Effect. | | |
| Table 3–1 | Schedule of Study Procedures and Assessments | 20 |
| Table 6–1 | Primary Objective(s) | 25 |
| Table 6–2 | Secondary Objective(s) | 25 |
| Table 6–4 | Safety Objective(s) | 26 |
| Table 9–1 | Test Product | 31 |
| Table 9–2 | Control Product | 34 |
| | List of Figures | |
| Figure 7-1 | Flowchart of Study Visits | 27 |
| Figure 11–1 | Categorization of All AEs | 45 |
| Figure 11–2 | Categorization of All SAE | 46 |

Status: Effective 

# 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to |
|---|---|
| | as soft contact lenses or contact lenses |
| Name of Control Product(s) | CooperVision® BIOFINITY® (comfilcon A) soft contact |
| Name of Control Floduct(s) | i i |
| | lenses (Biofinity contact lenses or Biofinity) |
| Adverse Device Effect | Adverse event related to the use of an investigational |
| (ADE) | medical device (test product) or control product. Note: This |
| | definition includes adverse events resulting from insufficient |
| | or inadequate instructions for use, deployment, |
| | implantation, installation, or operation; any malfunction; |
| | and use error or intentional misuse of the test product or |
| | control product. |
| Advorgo Event (AE) | Any untoward medical occurrence, unintended disease or |
| Adverse Event (AE) | |
| | injury, or untoward clinical signs (including abnormal |
| | laboratory findings) in subjects, users or other persons, |
| | whether or not related to the investigational medical device |
| | (test product). Note: For subjects, this definition includes |
| | events related to the test product, the control product, or the |
| | procedures involved. For users or other persons, this |
| | definition is restricted to events related to the test product. |
| | Requirements for reporting Adverse Events in the study can |
| | be found in Section 11. |
| Anticipated Cariava | Cariava advana davias affast which havita natura in illustra |
| Adversa Davisa Effect | Serious adverse device effect which by its nature, incidence, |
| Adverse Device Effect | severity, or outcome has been identified in the risk |
| | management file. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, |
| | quality, durability, reliability, safety, or performance. Note: |
| | This definition includes malfunctions, use errors, and |
| | inadequate labeling. |

Document: TDOC-0057524

Version: 1.0; CURRENT; Most-Recent; Effective Status: Effective 

| | Requirements for reporting Device Deficiencies in the study |
|---|---|
| | can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for |
| | participation in the study. |
| Interventional Clinical Trial | A research trial that prospectively assigns, whether |
| | randomly or not, human participants or groups of humans to |
| | one or more health-related interventions to evaluate the |
| | effects on health outcomes, and/or a research trial in which |
| | diagnostic or monitoring procedures beyond standard of care |
| | are conducted and generate outcomes for use in analysis of |
| | _ |
| | data. |
| Investigational Product (IP) | Is defined as a preventative (vaccine), a therapeutic (drug or |
| investigational Froduct (if ) | biologic), device, diagnostic, or palliative used as a test or |
| | control product in a clinical trial, including a product with a |
| | marketing authorization when used or assembled |
| | (formulated or packaged) in a way different from the |
| | authorized form, or when used for an unauthorized |
| | indication, or when used to gain further information about |
| | the authorized form. |
| Malfunction | Failure of a medical device to perform in accordance with its |
| | intended purpose when used in accordance with the |
| | instructions for use or clinical investigation plan. |
| Non-serious Adverse Event | Adverse event that does not meet the criteria for a serious |
| | adverse event. |
| Randomized Subjects | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| Serious Adverse Event | Adverse event that led to any of the following: |
| (SAE) | D. d |
| | • Death. |

Status: Effective 

• A serious deterioration in the health of the subject that either resulted in:

- a. a life-threatening illness or injury.

  Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form.
- b. any potentially sight-threatening event or permanent impairment to a body structure or a body function.
- c. in-patient hospitalization or prolonged hospitalization.

*Note: Planned hospitalization for a pre*existing condition, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

- d. a medical or surgical intervention to preventa) or b).
- e. any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.

Document: TDOC-0057524 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

| | Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 11 for additional SAEs. |
|---|---|
| Significant Non-Serious<br>Adverse Event | Is a symptomatic, device-related, non-sight threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. |
| | Refer to Section 11 for additional Significant Non-Serious AEs. |
| Unanticipated Serious Adverse Device Effect | Serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the risk management file. |
| Use Error | Act or omission of an act that results in a different medical device response than intended by manufacturer or expected by user. Note: This definition includes slips, lapses, and mistakes. An unexpected physiological response of the subject does not in itself constitute a use error. |

Status: Effective 

## 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2-1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| Biofinity contact | CooperVision BIOFINITY (comfilcon A) soft contact lenses |
| lens or Biofinity | (LID010221) |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CLCDVA | Contact lens corrected distance visual acuity |
| CLEAR CARE | CLEAR CARE® Cleaning & Disinfecting Solution |
| CRF | Case report form |
| D | Diopter(s) |
| D/C | Discontinue |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FAS | Full analysis set |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| IEC | |
| IEC | Independent ethics committee |
| IP | Investigational and dust |
| IRB | Investigational product Institutional review board |
| ISO | International Organization for Standardization |
| 150 | International Organization for Standardization |
| LID | Lens identification |
| logMAR | Logarithm of the minimum angle of resolution |
| contact | soft contact lenses (LID018869) |
| lens or | soft contact lenses (LiDo18889) |
| N/A | Not applicable |
| OD | Right eye |


Status: Effective 

| Abbreviation | Definition |
|--------------|------------------------------------|
| OS | Left eye |
| OU | Both eyes |
| PP | Per protocol analysis set |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SiHy | Silicone hydrogel |
| SOP | Standard operating procedure |
| UCDVA | Uncorrected distance visual acuity |
| US / USA | United States of America |
| USV | Unscheduled visit |
| VA | Visual acuity |
| VS | Versus |

Status: Effective 

#### 3 PROTOCOL SUMMARY

| This will be a prospective, randomized, | | controlled, double- |
|------------------------------------------|------------|---------------------|
| masked, parallel-group daily wear clinic | cal study. | |

Approximately 16 sites in the US will enroll approximately 160 subjects. Subjects will be expected to attend 4 office visits: Screening/Baseline/Dispense, Week 1 Follow-up, Month 1 Follow-up, and Month 3 Follow-up/Exit. The total expected duration of participation for each subject is approximately 3-4 months in this daily wear clinical study. Accounting for both screen failure and dropout rates, approximately 96 subjects will be assigned to wear the test lenses and 48 subjects will be assigned to wear the control lenses,

| lenses and 40 subjects will be assigned to wear the control lenses, | |
|---|---|
| | _ |

Subjects and the study personnel conducting the study evaluations will be masked to treatment. Subjects who meet the inclusion and exclusion criteria will be randomized to wear either the test contact lenses in both eyes or the control contact lenses (Biofinity) in both eyes for 3 months of daily wear exposure.



At the Screening/Baseline/Dispense Visit, study lenses will be dispensed to qualified subjects

| Alcon - Business Use O | <sub>-</sub> ) | <b>)ate:</b> 26-May-2020 |
|---|---|---|
| <b>Document:</b> TDOC-0057524 <b>Status:</b> Effective | Version: 1.0; CURRENT; Most-Recent; Effective | Page <b>14</b> of <b>62</b> |
| | All study lenses will be worn for at least 5 days pe | r week and |
| 8 hours per day in a daily | wear modality (eg, will not be worn while sleeping). | |
| . Rega | rdless of whether the subject is randomized to the test | or the control |
| group, CLEAR CARE C | leaning & Disinfecting Solution (CLEAR CARE) mus | st be used for |
| cleaning and disinfection | | |
| Investigational | Medical Device | |
| product type | | |
| Study type | Interventional | |
| Investigational | Test Product: soft contact lens | |
| products | Control Product: Biofinity soft contact lens | |
| Purpose and | The purpose of this clinical study is to evaluate the sa | fety and |
| rationale | performance of the investigational soft conta | ct lens |
| | compared to the commercially available Biofinity sof | t contact |
| | lens, when worn in a daily wear modality, by assessing | ıg visual |

Printed By: Print Date:

acuity as the primary endpoint.

Status: Effective 

| Objective(s) | The primary effectiveness objective is to demonstrate noninferiority of compared to Biofinity in CLCDVA at Week 1 Follow-up. The secondary effectiveness objective is to demonstrate noninferiority of compared to Biofinity in the percentage of subjects achieving CLCDVA 20/20 or better, in each eye, at Week 1 Follow-up. |
|---|---|
| Endpoint(s) | Primary Effectiveness • Mean contact lens corrected distance visual acuity (CLCDVA, Snellen converted to logMAR) in each eye at Week 1 Follow-up Secondary Effectiveness • Percentage of subjects achieving CLCDVA 20/20 or better in each eye, at Week 1 Follow-up |

Status: Effective 

# Safety

AEs

# Biomicroscopy findings Device deficiencies Effectiveness Assessment(s) VA with study lenses (Snellen distance)

Effective Date: 26-May-2020


Status: Effective 

| Study Design | Safety AEs Biomicroscopy Device deficiencies This will be a prospective, randomized, controlled, double-masked, parallel-group, daily wear clinical study. Subject participation in the study will be approximately 3 – 4 months with approximately 3 months of exposure to study lenses. |
|---|---|
| Subject population | Volunteer subjects aged 18 or over who are adapted daily wear |
| | frequent replacement soft contact lens wearers, excluding Biofinity habitual wearers, have at least 3 months of soft contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 8 hours per day. |
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day</li> <li>Manifest cylinder ≤ 0.75 D in each eye</li> </ul> |

Status: Effective 

| Status: Effective | | | Page 18 of 6 |
|---|---|---|---|
| | - | e corrected visual acuity | , , |
| | refraction) of | 20/20 or better in each | eye |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | modality (rou week) over the Monovision ( | tual contact lenses in an attinely sleeping in lenses are last 3 months prior to or multifocal contact lenses aring Biofinity lenses | s for at least 1 night per<br>enrollment |
| Data analysis | data from a pre-dete<br>from CLY935-C010 | ary and secondary effect<br>rmined subset of subject<br>will be combined with<br>will be performed on the | ets (see Section 12)<br>the current study, and |
| | Endpoint | Comparison | Statistical Method |
| | Primary | l | |
| | Mean CLCDVA<br>(Week 1<br>Follow-up) | vs Biofinity Noninferiority (margin = 0.10 logMAR) | Mixed effects<br>repeated measures<br>model |
| | Secondary | , | |
| | Proportion of subjects with CLCDVA of 20/20 or better in both eyes (Week 1 Follow-up) | vs Biofinity Noninferiority (margin = 0.10) | Generalized linear mixed model |
| | No inferential testin | g will be carried out for | safety endpoints. |

Status: Effective 



Table 3-1 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense Day 1 | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Month 1<br>Follow-up <sup>5</sup><br>Day 30 | Visit 4 Month 3 Follow-up/Exit <sup>5</sup> Day 95 | Early<br>Exit | usv |
|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | |
| Demographics | X | | | | | |
| Medical History | X | X | X | X | X | (X) |
| Pregnancy | X | X | X | X | X | (X) |
| Concomitant Medications | X | X | X | X | X | (X) |
| Inclusion/Exclusion | X | | | | | |
| Habitual lens information (brand/manufacturer, power, modality/wear success, habitual lens care brand) | X | | | | | |
| | | | | X | | |
| Biomicroscopy | X | X | X | X | X | (X) |
| Randomize and record lens power | X | | | | | |

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense Day 1 | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Month 1<br>Follow-up <sup>5</sup> | Visit 4 Month 3 Follow-up/Exit <sup>5</sup> Day 95 | Early<br>Exit | usv |
|---|---|---|---|---|---|---|
| IP Dispense* | X | (X) | X | | | (X) |
| VA w/ study lenses (OD, OS Snellen distance) | X | X | X | X | X | (X) |

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense Day 1 | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Month 1<br>Follow-up <sup>5</sup> | Visit 4 Month 3 Follow-up/Exit <sup>5</sup> Day 95 | Early<br>Exit | usv |
|---|---|---|---|---|---|---|
| Adverse Events | X | X | X | X | X | (X) |
| Device deficiencies | X | X | X | X | X | (X) |
| Exit Form | (X) | (X) | (X) | X | X | (X) |



| Alcon - Business Use Only Document: TDOC-0057524 | Protocol - Version: 1.0; | CURRENT; Most-Rece | | te: 26-May-2020 |
|---|---|---|---|---|
| Status: Effective | | | | |
| | | | | i |
| 5 INTRODUCTION | | | | |
| In this clinical study, the perfo<br>compared to the commercially | | | | |
| demonstrate the safety and eff | | | ens, both to be v | |
| daily wear modality and repla | | | | |
| for vision correction. Therefor | re, the measurem | ent of distance VA | is planned as th | ne primary |
| effectiveness variable. | | | | |




Status: Effective 



Refer to the IB for additional information.

## **6 STUDY OBJECTIVES**

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|------------------------------------|-----------------------------------|
| Demonstrate noninferiority of | Mean CLCDVA in each eye at Week 1 |
| compared to Biofinity in CLCDVA at | Follow-up. |
| Week 1 Follow-up. | |

# 6.2 Secondary Objective(s)

Table 6–2 Secondary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Demonstrate noninferiority of compared to Biofinity in the percentage of subjects achieving CLCDVA 20/20 or better in each eye, at Week 1 Follow-up. | Percentage of subjects achieving CLCDVA 20/20 or better in each eye at Week 1 Follow-up. |

Status: Effective 

# 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|-----------------------------------------------|------------------------|
| Duty of care and evaluation of safety profile | AEs |
| of the investigational products. | Biomicroscopy findings |
| | Device deficiencies |

| of the investigational products. | Biomicroscopy findings Device deficiencies |
|---|---|
| 7 INVESTIGATIONAL PLAN | N |
| 7.1 Study Design | |
| This will be a prospective, randomized masked, parallel-group, daily wear clin | |
| This clinical study will engage approxi<br>160 subjects with approximately 10 - 1 | imately 16 clinic sites to enroll approximately 5 subjects per site. |
| Follow-up, Month 1 Follow-up, and M participation for each subject is approx exposure to study lenses in this daily w | ffice visits: Screening/Baseline/Dispense, Week 1 fonth 3 Follow up/Exit. The total expected duration of timately 3-4 months with approximately 3 months of year study. Subjects will be randomized to wear either eyes or the control Biofinity contact lenses in both |
| Following randomization, study lenses | will be dispensed to the subject. |
| Subjects will wear the lenses while awaysed for daily cleaning and disinfection | ake in a daily wear modality. CLEAR CARE will be |

| Tone wing randomization, study renses win of dispensed to the subject |
|---|
| Subjects will wear the lenses while awake in a daily wear modality. CLEAR CARE will be |
| used for daily cleaning and disinfection. |

Status: Effective 

Figure 7-1 Flowchart of Study Visits



## 7.4 Rationale for Choice of Control Product

The Biofinity contact lens was chosen as the control product because this lens is a proper predicate device to compare to contact lens with regard to effectiveness and safety. Both the contact lens and Biofinity contact lens are frequent replacement SiHy lenses and are to be prescribed for daily wear. The Biofinity contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes. The lenses are intended to be cleaned and disinfected daily when worn for daily wear.

Status: Effective 

#### **8 STUDY POPULATION**

The study population consists of adult male or female subjects (aged 18 or over), with non-diseased eyes, who require optical correction for refractive ametropia

The intended study population consists of volunteer subjects who are frequent replacement daily wear soft contact lens wearers, excluding Biofinity habitual wearers, who have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and 8 hours per day.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill **all** of the following criteria:

- 1. At least 18 years of age.
- 2. Able to understand and sign an IRB/IEC approved Informed Consent form.
- 3. Willing and able to attend all scheduled study visits as required per protocol.
- 4. Successful wear of frequent replacement spherical daily wear soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
- 5. Manifest cylinder  $\leq 0.75$  D in each eye.

Alcon - Business Use Only Protocol - Effective Date: 26-May-2020
6. Best spectacle corrected (using manifest refraction) VA 20/20 or better in each eye.

## 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

| _ |
|---|
| _ |

Status: Effective 



Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation.

# 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

## 9 TREATMENTS ADMINISTERED

## 9.1 Investigational Product(s)

Test Product(s): soft contact lenses

Control Product(s) (If applicable): Biofinity (comfilcon A) soft contact lenses

Table 9–1 Test Product

| Test Product | soft contact lenses ( contact lens) (LID018869) |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended purpose in the current study | The intended use of this contact lens is for vision correction. |



Status: Effective  Usage Wear: o Daily Wear During waking hours only. o Bilateral Exposure: At least ~8 hours per day and ~5 days per week over a ~3-month exposure period. Lens Care: CLEAR CARE (mandatory), Packaging Blister foil pack description


Status: Effective  Storage conditions Stored at room temperature.


Status: Effective 

## **Table 9–2** Control Product

| Control Product(s) | Biofinity (comfilcon A) soft contact lenses (Biofinity contact lens) (LID010221) |
|---|---|
| Manufacturer | CooperVision |
| Indication for Use | The intended use of this contact lens is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: comfilcon A</li> <li>Water content: 48%</li> <li>Base curve: 8.6 mm</li> <li>Diameter: 14.0 mm</li> </ul> |
| Formulation | Silicone Hydrogel. Additional details can be found in the Biofinity package insert. |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>During waking hours only.</li> </ul> </li> <li>Bilateral</li> <li>Exposure: At least ~8 hours per day and ~5 days per week over a ~3-month exposure period.</li> </ul> |


Status: Effective 

| Number/Amount of Product to be Provided to the subject Packaging description Storage conditions Stored at room temperature. | Status: Effective | Page <b>35</b> of <b>62</b> |
|---|---|---|
| Product to be Provided to the subject Packaging description Blister foil pack. | | • |
| Provided to the subject Packaging description Blister foil pack. | Number/Amount of | |
| subject Packaging description Blister foil pack. | Product to be | lenses to last until the next planned study visit, allowing for planned |
| description | | and unplanned lens replacements. |
| | | Blister foil pack. |
| Storage conditions Stored at room temperature. | description | |
| Storage conditions Stored at room temperature. | | |
| · | Storage conditions | Stored at room temperature. |

or Biofinity

Printed By: Print Date:

Subjects will be randomized in a 2:1 manner to receive either the

contact lenses, respectively.




It is the Investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- •
- All unused products are available for return to the Study Sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related AE
  (ie, ADE or SADE) are returned to the Study Sponsor for investigation, unless
  otherwise directed by the Sponsor.

The Investigator is responsible for proper disposition of all unused IPs at the conclusion of the study.

# 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the Investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned


Status: Effective 

• Any non-drug therapies (including physical therapy and blood transfusions).

The Investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 4 office visits, as shown below.

| Visit # | Visit Type | Visit Day |
|---------|------------------------------|-----------|
| Visit 1 | Screening/Baseline/Dispense | Day 1 |
| Visit 2 | Week 1 Follow-up Visit | Day 8 |
| Visit 3 | Month 1 Follow-up Visit | Day 30 |
| Visit 4 | Month 3 Follow-up/Exit Visit | Day 95 |

Unscheduled Visits and Early Termination Visits are allowed, if necessary.



At the Screening/Baseline/Dispense Visit, study lenses will be dispensed to the subject. All subjects will wear the study lenses in a daily wear modality, only during waking hours.



Status: Effective 

### 10.1 Informed Consent and Screening

The Investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

The Investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

### **10.2 Description of Study Procedures and Assessments**

# 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

# **10.2.2** Medical History and Concomitant Medications

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

# **10.2.3** Investigational Product compliance

Review subject compliance with the IP usage

Status: Effective 

### 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit. Requirements for reporting AEs in the study can be found in Section 11.

### 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment

Slit-lamp examination of the cornea, iris/anterior chamber, and lens must be performed in both eyes before instillation of any diagnostic eye drops.

Slit-lamp examination of the tear film stability will also be performed at each visit.

### 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11.



# 10.5 Discontinued Subjects

#### 10.5.1 Screen Failures

Screen failures are subjects who were excluded from the study after signing the informed consent, not meeting the inclusion/exclusion criteria, and prior to randomization to product/dispense of study product.

The Investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.


Status: Effective 

#### 10.5.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the Investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be re-used.

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the Investigator, continued treatment poses a risk to their health.



# **10.6 Clinical Study Termination**

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

- The Study Sponsor must:
  - o Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
  - o Inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.

Status: Effective 

The Investigator must:

- Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
- Provide subjects with recommendations for post-study treatment options as needed.

The Investigator may terminate the site's participation in the study for reasonable cause.

### 10.6.1 Follow-up of subjects after study participation has ended

Study visits are not a substitute for routine eye care. Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test article). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11–1 Categorization of All AEs



Status: Effective 

Figure 11-2 Categorization of All SAE



#### **SAEs**

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the Investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics\*:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification


Status: Effective 

- Hypopyon
- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

#### Significant Non-Serious AE

A significant non-serious AE is a device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the Investigator must report any occurrence of the following as a Significant Non-Serious Adverse Event:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to Grade 3
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that persists for 2 or more weeks
- Neovascularization score greater than or equal to Grade 2

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with subject harm (ie, ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The Investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any subject harm separately.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the Investigator must document all device deficiencies reported or observed with test and control products on the Device Deficiency eCRF.


Status: Effective 

 ADEs or SAEs are documented on the Serious Adverse Event and Adverse Device Effect eCRF within 24 hours of the Investigator's or site's awareness.

- Device deficiencies are documented on the *Device Deficiency* eCRF within 24 hours of the Investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
   Certificate of Death, etc, if applicable, in narrative section of the Serious Adverse
   Event and Adverse Device Effect eCRF.

#### **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based upon medical judgment with consideration of any subjective symptom(s), as defined below:


Status: Effective 

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).

| Document: TDOC-0057524 Version: 1.0; CURRENT; Most-Recent; Effective Page 51 or | f <b>62</b> |
|---|---|
| 11.5 Unmasking of the Study Treatment | |
| Masked information on the identity of the assigned medical device should not be disclosed during the study. | |
| 11.6 Follow-Up of Subjects with AEs | |
| The Investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study. | : |
| | _ |
| | _ |
| 11.7 Pregnancy in the Clinical Study | |
| Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. | <b>)</b> |

Effective Date: 26-May-2020

Alcon - Business Use Only Protocol -

Status: Effective 

#### 12 ANALYSIS PLAN

lenses evaluated in this study,

Printed By:

post-baseline (post-Dispense) CLCDVA.

Data from a subset of subjects in the CLY935-C010 study will be combined with data from this study. This combined set will serve as the basis for all planned analyses for the primary and secondary effectiveness objectives. Subjects in CLY935-C010 will be included in the combined set only if they satisfy the following criterion:

| and secondary effectiveness objectives. Subjects in CLY935-C010 will be included in the combined set only if they satisfy the following criterion: |
|---|
| • BCVA of 20/20 or better in each eye at the Screening/Baseline/Dispense Visit |
| · |
| 12.1 Subject Evaluability |
| Final subject evaluability must be determined prior to breaking the code for masked treatment (lens) assignment and locking the database, |
| 12.2 Analysis Sets |
| 12.2.1 Safety Analysis Set |
| Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, For treatment-emergent safety analyses, subjects/eyes will be categorized |
| under the actual study lenses exposed. |
| 12.2.2 Full Analysis Set |

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study

Print Date:

, and who have at least one


Status: Effective 

## 12.2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the DEP.

### 12.3 Demographic and Baseline Characteristics

Demographic information, recent lens-wearing experience (including wear modality and wear success), and habitual lens information will be presented by lens group and overall. Counts and percentages will be presented for categorical variables such as sex, age group, race, an ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

## 12.4 Effectiveness Analyses



# 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary effectiveness objective is to demonstrate noninferiority of compared to Biofinity in mean CLCDVA at Week 1 Follow-up.

The primary endpoint is the mean CLCDVA at Week 1 Follow-up. The corresponding assessment is collected with study lenses, in Snellen, for each eye. Conversion will be made to the logMAR scale.

# 12.4.1.1 Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.10 (in logMAR scale) for noninferiority:

H<sub>0</sub>: 
$$\mu_{(T)} - \mu_{(C)} \ge 0.10$$
  
H<sub>a</sub>:  $\mu_{(T)} - \mu_{(C)} < 0.10$ 


Status: Effective 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the Week 1 Follow-up mean CLCDVA for contact lenses, respectively, on the logMAR scale.

### 12.4.1.2 Analysis Methods

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, visit (Dispense, Week 1 Follow-up, Month 1 Follow-up, and Month 3 Follow-up), and lens-by-visit interaction as fixed effects.

Within-subject correlation due to eye will also be accounted for in the model. Lens difference (minus Biofinity) and the corresponding two-sided 95% CI will be computed for 1-Week Follow-up. Noninferiority in CLCDVA will be declared if the upper confidence limit is less than 0.10.

# 12.4.2 Analysis of Secondary Effectiveness Endpoints

The secondary effectiveness objective is to demonstrate noninferiority of compared to Biofinity in the percentage of subjects achieving distance VA 20/20 or better, in each eye, at Week 1 Follow-up.

The corresponding endpoint is the percentage (proportion) of subjects with CLCDVA of 20/20 or better, measured monocularly, in both OD and OS at Week 1 Follow-up.

# **12.4.2.1** Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.10 (10%) for noninferiority.

$$H_0$$
:  $P_{(T)} - P_{(C)} \le -0.10$   
 $H_a$ :  $P_{(T)} - P_{(C)} > -0.10$ 

where  $P_{(T)}$  and  $P_{(C)}$  denote the proportion of subjects attaining at least 20/20 in CLCDVA at Week 1 Follow-up in each eye (OD and OS) for and Biofinity contact lenses, respectively.

# 12.4.2.2 Analysis Methods

A binary variable will be defined for each subject to indicate whether the CLCDVA at Week 1 Follow-up is no worse than 20/20 in both OD and OS, and the corresponding proportion will be computed for each lens using the number of subjects as the denominator.

. From the two-sided 95% CI on the lens difference ( minus Biofinity),


Status: Effective 

noninferiority in proportion of subjects achieving 20/20 or better in CLCDVA in both eyes will be declared if the lower confidence limit is greater than -0.10.

| <u> </u> |
|----------|

| Alcon - Business Use Uniy Pa | rotocol - | ate: 20-May-2020 |
|---|---|---|
| Status: Effective | | Page <b>56</b> of <b>62</b> |

## 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy Findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of AE as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation, significant non-serious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Two listings for device deficiencies, prior to exposure of study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated. No inferential testing will be done for safety analysis. 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS 13.1 Subject Confidentiality The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant.

Version: 1.0; CURRENT; Most-Recent; Effective

Alcon - Business Use Only Protocol -

Document: TDOC-0057524

Status: Effective

Effective Date: 26-May-2020




# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the Study Sponsor and are independent of study site staff.



#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

### 13.4 Sponsor and Monitoring Responsibilities

The Study Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate Study Sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

A Coordinating Investigator may be identified by the Study Sponsor to review and endorse the final study report. In cases where a Coordinating Investigator is engaged, the Study Sponsor will select the Coordinating Investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

Status: Effective 

### 13.5 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Study Sponsor and the Investigator's files will be reviewed as part of the ongoing study monitoring.

### 13.6 Quality Assurance and Quality Control

The Study Sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the Study Sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the Study Sponsor with the Investigator/Institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS



The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed,



The Study Sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov as required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be

Alcon - Business Use Only Protocol - Effective Date: 26-May-2020 Document: TDOC-0057524 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

made publicly available on www.clinicaltrials.gov regardless of outcome as required by current regulations and, if applicable, in other public databases as required by local country regulations.

| _ |
|---|
| _ |

Alcon - Business Use Only Protocol - Effective

Document: TDOC-0057524 Version: 1.0; CURRENT; Most-Recent; Effective Effective Date: 26-May-2020

Status: Effective

# Signature Page for V-CLN-0000052 v1.0



Signature Page for V-CLN-0000052 v1.0